CLINICAL TRIAL: NCT01403220
Title: The Efficacity of Hemodiafiltration Versus Hemofiltration for Renal Insufficiency During Intensive Care: a Randomized, Open, Cross-over Study
Brief Title: The Efficacity of Hemodiafiltration Versus Hemofiltration for Renal Insufficiency During Intensive Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LOCAL/2011/PJ-02; 2011-A01550-41 (Other: ANSM)
Record Dates: First submitted 2011-07-25; First posted 2011-07-27 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2015-03

CONDITIONS: Renal Failure, Acute
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (hemodiafiltration first) (Active Comparator): This group of patients will alternate consecutive dialysis sequences between hemodiafiltration and hemofiltration, but starting with hemodiafiltration.
  Interventions: Procedure: Hemodiafiltration first
- Group 2 (hemofiltration first) (Active Comparator): This group of patients will alternate consecutive dialysis sequences between hemodiafiltration and hemofiltration, but starting with hemofiltration.
  Interventions: Procedure: Hemofiltration first

INTERVENTIONS:
Procedure: Hemodiafiltration first — Patients will alternate consecutive dialysis sequences between hemodiafiltration and hemofiltration, but starting with hemodiafiltration.
  Arms: Group 1 (hemodiafiltration first)
Procedure: Hemofiltration first — Patients will alternate consecutive dialysis sequences between hemodiafiltration and hemofiltration, but starting with hemofiltration.
  Arms: Group 2 (hemofiltration first)

SUMMARY:
The primary objective of this study is to compare the efficacity of hemodiafiltration and hemofiltration for decreasing plasma urea at 12h among intensive care patients. Secondary objectives include comparing urea clearance, filter duration, and %down-time, between the two techniques.

ELIGIBILITY:
Inclusion Criteria:

* According to RIFLE score, patient is stage 'F'
* The patient must be insured or beneficiary of a health insurance plan
* The patient meets at least one of the following criteria:
* metabolic acidosis (pH < 7.2), excluding keto-acidosis
* plasma urea > 25 mmol/l
* hyper-hydration is not controlled by diuretics

Exclusion Criteria:

* Chronic, terminal renal insufficiency with dialysis
* The patient is under judicial protection, under tutorship or curatorship
* Suspect hyperkaliemia (Kaliemia > 6.5 mmol/l with electrocardiographic effects)
* Intoxications treated via dialysis
* Pregnant, lactating, parturient women
* Medical indication for localized citrate anticoagulation
* dialysis of less than 12 h
* patient or representative refuses to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2012-04; Primary Completion 2015-03-17 (Actual); Study Completion 2015-03-17 (Actual)

PRIMARY OUTCOMES:
Proportion of dialysis sequences for which the rate of plasma urea reduction > 60%. | 12 hours
  Proportion of dialysis sequences for which the rate of plasma urea reduction > 60%. Rate of plasma urea reduction = (initial urea concentration - urea concentration after 12h our dialysis)/initial urea concentration.

SECONDARY OUTCOMES:
Proportion of dialysis sequences for which the rate of plasma urea reduction > 60%. | 24 hours
  Proportion of dialysis sequences for which the rate of plasma urea reduction > 60%. Rate of plasma urea reduction = (initial urea concentration - urea concentration after 12h our dialysis)/initial urea concentration.
Urea clearance (ml/min) for the dialysis sequence under study | 12 hours
  Urea clearance (ml/min) for the dialysis sequence under study.
Filter lifespan (hours) for the dialysis sequence under study. | 12 hours.
  Filter lifespan (hours) for the dialysis sequence under study.
The percentage down-time for the first 24 hours of dialysis | 24 hours
  The percentage down-time for the first 24 hours of dialysis = (number of hours where the exchange is not effective / 24 hours)*100
Fluid replacement (yes/no) | 12 hours
  Was fluid replacement necessary during the studied dialysis sequence?
Fluid replacement (yes/no) | 24 hours
  Was fluid replacement necessary during the studied dialysis sequence?

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Jeannes, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- Centre Hospitalier Universitaire de Nîmes, Nîmes, Gard, France

REFERENCES:
- [Result] Roger C, Muller L, Wallis SC, Louart B, Saissi G, Lipman J, Lefrant JY, Roberts JA. Population pharmacokinetics of linezolid in critically ill patients on renal replacement therapy: comparison of equal doses in continuous venovenous haemofiltration and continuous venovenous haemodiafiltration. J Antimicrob Chemother. 2016 Feb;71(2):464-70. doi: 10.1093/jac/dkv349. Epub 2015 Nov 3. PMID 26538503
- [Derived] Roger C, Wallis SC, Muller L, Saissi G, Lipman J, Bruggemann RJ, Lefrant JY, Roberts JA. Caspofungin Population Pharmacokinetics in Critically Ill Patients Undergoing Continuous Veno-Venous Haemofiltration or Haemodiafiltration. Clin Pharmacokinet. 2017 Sep;56(9):1057-1068. doi: 10.1007/s40262-016-0495-z. PMID 28035589
- [Derived] Roger C, Wallis SC, Muller L, Saissi G, Lipman J, Lefrant JY, Roberts JA. Influence of Renal Replacement Modalities on Amikacin Population Pharmacokinetics in Critically Ill Patients on Continuous Renal Replacement Therapy. Antimicrob Agents Chemother. 2016 Jul 22;60(8):4901-9. doi: 10.1128/AAC.00828-16. Print 2016 Aug. PMID 27270279